CLINICAL TRIAL: NCT05471037
Title: Swiss Multicenter Randomized Controlled Trial on Different Limb Lengths in Gastric Bypass Surgery (SLIM Trial) - Part 3: Metabolic Mechanisms and Inflammatory Response
Brief Title: Different Limb Lengths in Gastric Bypass Surgery (SLIM) - Part 3: Metabolism and Inflammation
Acronym: SLIM - Part 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SLIM - Part 3
Record Dates: First submitted 2022-03-21; First posted 2022-07-22 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Long Biliopancreatic Limb LRYGB (Active Comparator): 25 morbidly obese patients undergoing gastric bypass surgery, participating in SLIM Trial.
  Interventions: Procedure: Long Biliopancreatic Limb LRYGB
- Short Biliopancreatic Limb LRYGB (Active Comparator): 25 morbidly obese patients undergoing gastric bypass surgery, participating in SLIM Trial.
  Interventions: Procedure: Short Biliopancreatic Limb LRYGB
- Control (No Intervention): 15 normal weight control group without surgery.

INTERVENTIONS:
Procedure: Long Biliopancreatic Limb LRYGB — LRYGB with an 180 cm biliopancreatic limb (BPL) and an alimentary limb (AL) of 80 cm.
  Arms: Long Biliopancreatic Limb LRYGB
Procedure: Short Biliopancreatic Limb LRYGB — Standard LRYGB with a 80 cm BPL and a 180 cm long AL.
  Arms: Short Biliopancreatic Limb LRYGB

SUMMARY:
Investigation of underlying metabolic mechanisms and impact on the two surgical procedures on inflammatory factors.

DETAILED DESCRIPTION:
The aim of this project is to investigate underlying metabolic mechanisms in a subpopulation of patients of the SLIM trial, where a laparoscopic proximal Roux-en-Y gastric bypass (LRYGB) with a longer biliopancreatic limb (BPL) is compared to a standard LRYGB. For this purpose, the aim is to examine differences in number of intestinal enteroendocrine cells, subpopulations of intestinal macrophages, and gene expression or DNA-methylation in tissue samples obtained by colonoscopy from the ileum and transverse colon. In addition, gut microbiota (from colon biopsy and fecal samples), meal-stimulated gut hormone profiles, glycemic control, and metabolite patterns (metabolomics; in blood, urine, stool and breath) including plasma bile acid concentrations preoperatively and 6 months post-surgery will be examined. Body composition (fat mass and lean mass) will be measured by means of BIA (bioimpedance analysis; Biacorpus).

ELIGIBILITY:
Inclusion Criteria:

* 2 x 25 patients with morbid obestiy (BMI of 35 kg/m2 or higher) who comply with the regulatory rules for bariatric surgery in Switzerland (SMOB guidelines) and participate in the SLIM Trial
* 15 healthy lean controls

Exclusion Criteria:

* general contraindications to kind of surgery
* known or suspected non-compliance
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders etc. of the participant
* participation in another interventional study
* BMI > 60 kg/m2
* height < 145 cm
* CL length of < 180 cm as measured intraoperatively
* ASA physical status classification > III
* inflammatory bowel disease
* diabetes
* intake of corticosteroids, anti-inflammatory/ immunosuppressive drugs potentially altering immune cells
* clinical signs of current infection
* known anemia (e.g. hemoglobin < 110g/L for males, < 100g/L for females)
* known neutropenia (e.g. leucocyte count < 1.5 x 10^9/L or ANC < 0.5 x 10^9/L)
* known immunodeficiency, e.g. HIV
* known vasculitis, collagenosis
* known adrenal insufficiency and/or substitution with glucocorticoids
* risky daily alcohol consumption (> 24g/d for males, > 12g/d for females)
* drug abuse
* known liver cirrhosis Child B or C
* known uncontrolled congestive heart failure
* known uncontrolled malignant disease
* currently pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in glucose tolerance | pre-OP and 6-8 months post-OP
  Change in glucose tolerance as measured by plasma glucose concentrations at 120 minutes after ingestion of a standardized liquid test meal, pre-OP and 6-8 months post-OP.

SECONDARY OUTCOMES:
glycemic control | pre-OP and 6-8 months post-OP
  Change in glucose variability measured by continuous glucose measurement over 1 week, pre-OP and 6-8 months post-OP.
intestinal glucose absorption rate | pre-OP and 6-8 months post-OP
  Differences in intestinal glucose absorption rate after ingestion of a standardized liquid test meal measured by 3-OMG
gastrointestinal peptides | pre-OP and 6-8 months post-OP
  Differences in the release of gastrointestinal peptides after ingestion of a standardized liquid test meal
intestinal enteroendocrine cells | pre-OP and 6-8 months post-OP
  Differences in number and phenotype (protein expression) of intestinal enteroendocrine cells (from ileum biopsies)
intestinal macrophages | pre-OP and 6-8 months post-OP
  Differences in the number and phenotype (gene expression, methylation) of intestinal macrophages and subpopulations (from colon biopsies)
gut microbiota composition | pre-OP and 6-8 months post-OP
  Differences in gut microbiota composition (from colon biopsy and fecal sample)
bile acids | pre-OP and 6-8 months post-OP
  Differences in bile acids and metabolomic patterns (blood)
inflammatory profile | pre-OP and 6-8 months post-OP
  Differences in inflammatory profile measured by hsCRP in blood
enterocyte gene expression | pre-OP and 6-8 months post-OP
  Differences in enterocyte gene expression or DNA-methylation (tissue samples from ileum biopsies)
appetite-related sensations | pre-OP and 6-8 months post-OP
  Differences in subjective appetite-related sensations (feelings of hunger, prospective food consumption, satiation and fullness) after liquid test meal, assessed with Visual Analog Scales
body composition | pre-OP and 6-8 months post-OP
  Body composition (measured by Bio Impedance Analysis (BIA))
mineral metabolism (blood) 1 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (creatinine) in blood samples.
mineral metabolism (blood) 2 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (phosphate) in blood samples.
mineral metabolism (blood) 3 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (calcium) in blood samples.
mineral metabolism (blood) 4 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (magnesium) in blood samples.
mineral metabolism (blood) 5 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (parathyroid hormone) in blood samples.
mineral metabolism (blood) 6 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (calcidiol) in blood samples.
mineral metabolism (blood) 7 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (calcitriol) in blood samples.
mineral metabolism (blood) 8 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (FGF23) in blood samples.
mineral metabolism (blood) 9 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (desoxypyridinoline) in blood samples.
mineral metabolism (blood) 10 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (bone alkaline phosphatase (bALP)) in blood samples.
mineral metabolism (blood) 11 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (osteocalcin) in blood samples.
mineral metabolism (blood) 12 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (sclerostin) in blood samples.
mineral metabolism (blood) 13 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (P1NP) in blood samples.
mineral metabolism (blood) 14 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (CTX) in blood samples.
mineral metabolism (stool) 1 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (phosphate) in feces samples.
mineral metabolism (stool) 2 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (calcium) in feces samples.
mineral metabolism (stool) 3 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (magnesium) in feces samples.
mineral metabolism (urine) 1 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (creatinine) in urine samples.
mineral metabolism (urine) 2 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (phosphate) in urine samples.
mineral metabolism (urine) 3 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (calcium) in urine samples.
mineral metabolism (urine) 4 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (magnesium) in urine samples.
mineral metabolism (urine) 5 | pre-OP and 6-8 months post-OP
  Differences in mineral metabolism parameter (desoxypyridinoline) in urine samples.
metabolomic patterns | pre-OP and 6-8 months post-OP
  Differences in metabolomic patterns assed in blood sample, urine sample, stool sample and exhaled breath.
immune response | pre-OP and 6-8 months post-OP
  Differences in immune response biomarkers in blood measured by a cytokine screening assay

CONTACTS AND LOCATIONS:
Overall Officials: Anne Christin Meyer-Gerspach, PD Dr. phil. II Dr. habil., Principal Investigator — St. Clara Forschung AG / St. Claraspital AG; Bettina Wölnerhanssen, PD Dr. med., Principal Investigator — St. Clara Forschung AG / St. Claraspital AG
Locations (1):
- St Clara Research Ltd, St Claraspital Basel, Basel, Switzerland